CLINICAL TRIAL: NCT00463905
Title: Evaluation of the Impact of a Case-finding Strategy for Vertebral Fractures on Bisphosphonate and Other Drug Prescribing in Primary Care, Using the Cohort for Skeletal Health in Bristol and Avon (COSHIBA)
Brief Title: Evaluation of the Impact of a Case-finding Strategy for Vertebral Fractures
Acronym: COSHIBA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Bristol (Other)
Responsible Party: Principal Investigator, Emma Clark, Consultant Senior Lecturer, University of Bristol
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Screening
Other Study IDs: SMED RJ4783
Record Dates: First submitted 2007-04-18; First posted 2007-04-20 (Estimated); Last update posted 2014-12-04 (Estimated); Status verified 2014-12

CONDITIONS: Osteoporosis; Vertebral Fracture
Keywords: osteoporosis; vertebral fractures; randomised controlled trial; screening
MeSH Terms: conditions — Osteoporosis; Spinal Fractures

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (No Intervention): Current management for identifying postmenopausal women with osteoporotic vertebral fractures in primary care i.e. nothing
- 2 (Experimental): Intervention arm: simple clinical assessment to identify high risk 30% (approximately) who will then be offered lateral thoraco-lumbar X-rays
  Interventions: Procedure: Clinical assessment +/- radiography

INTERVENTIONS:
Procedure: Clinical assessment +/- radiography — Clinical assessment: height loss, history of fracture, Margolis pain score, rib/pelvis distance
  Arms: 2

SUMMARY:
Postmenopausal women with vertebral fractures (VFs) represent an important target for secondary fracture prevention, but few of these patients come for clinical attention. Recent evidence suggests that screening postmenopausal women for clinical risk factors like height loss and fracture risk identifies those at high risk of prevalent VFs who should be referred for diagnostic X-rays, a strategy which is likely to prove cost effective. However, before being applied at a United Kingdom (UK)-wide level, it needs to be established that use of this strategy improves secondary fracture prevention, and that these benefits are achieved in a cost-effective manner. To examine these questions, a randomised-controlled-trial will be performed in which women aged 65-80 from general practitioner (GP)-practices in the intervention group will be invited for risk factor assessment, followed by referral for thoracolumbar X-ray where appropriate. The primary outcome will be a change in bisphosphonate or other drug prescribing between the intervention and control arms after six months.

DETAILED DESCRIPTION:
This study will use a randomised controlled trial to assess the impact of a case-finding strategy for vertebral fractures on bisphosphonate and other drug prescribing in primary care. A sample of postmenopausal women aged 65-80 years from Bristol will be invited to take part. They will be individually randomised into either the intervention or control arm in a 2:1 ratio in favour of controls. The participants in the intervention arm will attend their GP practice to receive a simple 15 minute assessment, and if found to be at high risk of vertebral fractures will have a thoracolumbar X-ray; those randomised to the control arm will receive current standard methods used to identify women at high risk of vertebral fractures (no active intervention). Follow-up will be for three years.

Baseline measurements will be taken from women in each arm via self-completion postal questionnaire, including current prescriptions of any bisphosphonate or other osteoporosis medication. The women in the intervention arm will attend their GP practice and receive a simple 15 minute assessment, and if found to be at high risk of vertebral fractures will have a thoracolumbar X-ray arranged for them. They will be given a leaflet on lifestyle interventions aimed to improve bone health. Women in the control arm will be sent the same leaflet. Post-intervention questionnaires will be sent to all women asking about fractures and current prescriptions of any bisphosphonate or other osteoporosis medication. The primary outcome will be the proportion of women prescribed medication for secondary fracture prevention in the intervention arm compared to the control arm. Secondary outcomes will include the proportion of fractures in the intervention versus control arm, and compliance with bisphosphonate or other drug prescribing.

This study will be performed subject to Research Ethics Committee (REC) approval, including any provisions of Site Specific Assessment (SSA), and local Research and Development approval. This study will be conducted in accordance with the Research Governance Framework for Health and Social Care and Good Clinical Practice.

ELIGIBILITY:
Inclusion Criteria:

* Female
* Aged 65-80 years
* Registered with a GP practice within Bristol Primary Care Trust (PCT)

Exclusion Criteria:

* None

Ages: 65 Years to 80 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 3200 (Actual)
Dates: Start 2007-10; Primary Completion 2009-06 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
The change in proportion of women aged 65-80 years prescribed bisphosphonates or other drugs in intervention arm compared with control arm | 2 years

SECONDARY OUTCOMES:
Number of extra VFs identified by risk-factor assessment tool | 2 years
Assessment of difference in indications for bisphosphonate prescribing after intervention | 2 years
Assessment of compliance | 2 years
Assessment of quality of life | 2 years
Economic analysis to assess cost-effectiveness of intervention | 2 years
Assessment of impact on fractures | 2 years
Assessment of whether algorithm based qualitative (ABQ) semi-quantitative method of analyzing X-rays is better than simple inspection in identifying vertebral fractures | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Emma M Clark, MBBS, PhD, Principal Investigator — University of Bristol
Locations (1):
- Bristol Primary Care Trust (PCT), Bristol, United Kingdom

REFERENCES:
- [Background] Clark EM, Gould VC, Morrison L, Masud T, Tobias J. Determinants of fracture risk in a UK-population-based cohort of older women: a cross-sectional analysis of the Cohort for Skeletal Health in Bristol and Avon (COSHIBA). Age Ageing. 2012 Jan;41(1):46-52. doi: 10.1093/ageing/afr132. Epub 2011 Nov 21. PMID 22107913
- [Background] Weston JM, Norris EV, Clark EM. The invisible disease: making sense of an osteoporosis diagnosis in older age. Qual Health Res. 2011 Dec;21(12):1692-704. doi: 10.1177/1049732311416825. Epub 2011 Aug 2. PMID 21810994
- [Result] Clark EM, Gould V, Morrison L, Ades AE, Dieppe P, Tobias JH. Randomized controlled trial of a primary care-based screening program to identify older women with prevalent osteoporotic vertebral fractures: Cohort for Skeletal Health in Bristol and Avon (COSHIBA). J Bone Miner Res. 2012 Mar;27(3):664-71. doi: 10.1002/jbmr.1478. PMID 22113935